CLINICAL TRIAL: NCT04059900
Title: A Double-blind, Randomised, Placebo-controlled Study on the Efficacy of Iberogast® (STW 5) in Patients With Functional Dyspepsia and Concomitant Reflux Symptoms Measured With Impedance and Wireless pH Monitoring
Brief Title: Study in Patients Suffering From Heartburn and Backward Flow of Stomach Liquid Into the Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20985; 2008-002305-40 (EudraCT Number)
Record Dates: First submitted 2019-07-12; First posted 2019-08-16 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — iberogast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STW5 (Iberogast®, BAY98-7411) (Experimental): The medication was applied daily per os (orally, p.o.) from day 0 to day 28. The dosage was 20 drops three times daily before the meals.
  Interventions: Drug: STW5 (Iberogast®, BAY98-7411)
- Placebo (Placebo Comparator): The medication was applied daily p.o. from day 0 to day 28. The dosage was 20 drops three times daily before the meals
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: STW5 (Iberogast®, BAY98-7411) — The medication was applied daily per os (orally, p.o.) from day 0 to day 28. The dosage was 20 drops three times daily before the meals.
  Arms: STW5 (Iberogast®, BAY98-7411)
Drug: Placebo — The medication was applied daily p.o. from day 0 to day 28. The dosage was 20 drops three times daily before the meals
  Arms: Placebo

SUMMARY:
In this study researchers want to learn more about the effectiveness of Iberogast® in patients with irritable stomach and concomitant chronic or recurrent heartburn and backward flow of stomach liquid into the esophagus. 60 patients in the age range from 18 - 80 year will be treated over 4 weeks with Iberogast® or placebo - an inactive substance which looks identical to Iberogast®. Patients completed diaries will provide researchers with detailed information on the change of stomach and intestinal symptoms during the treatment period. In addition information on the acidity of the esophagus and stomach liquid will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex aged 18-80 years.
2. Diagnosis of functional dyspepsia according to Rome III criteria:

   * Pain or burning localized to the epigastrium of at least moderate severity at least once per week with a total duration of at least 6 months.
   * Pain was intermittent.
   * Pain was not generalized or localized to other abdominal or chest regions.
   * Pain was not relieved by defecation or passage of flatus.
   * Pain did not fulfil criteria for gallbladder and sphincter of Oddi disorders.
3. At assessment (visit 1 or 3) three items of GIS had to be judged at least as moderate including reflux symptoms, but reflux symptoms not dominating the clinical picture.
4. Endoscopy of the upper gastrointestinal tract and abdominal sonography without pathological findings that could have explained the symptoms (findings of up to 5 gastric erosions could be tolerated if patient had no concomitant intake of acetylsalicylic acid).
5. Patients willing to comply with the study protocol.
6. Patients who were able to understand and provide written informed consent to participate in the trial (signed informed consent).

Exclusion Criteria:

1. Concomitant treatment during the study with any medication that could influence the gastrointestinal function (e.g. prokinetics, antacids, antibiotics, antidepressant, laxatives, calcium antagonists, beta-blocker, antidiarrheics).
2. Regular intake of nonsteroidal antiphlogistic drugs incl. cyclooxygenase-2 (COX-2)-inhibitors (exception: acetylsalicylic acid for cardiovascular prevention up to 100 mg daily).
3. History of clinically relevant gastrointestinal disease such as gastric-, pancreatic-, colon-, rectal-cancer.
4. History of gastric and/or duodenal ulcer.
5. History of abdominal surgery (cholecystectomy and appendectomy could be tolerated).
6. History and/or presence of coronary heart disease.
7. Known intolerance to azo dyes E 110 and E 151.
8. Food allergies and known lactose intolerance.
9. Evidence of any gastrointestinal infectious diseases.
10. Participation in a clinical trial 30 days prior to this trial.
11. Concurrent participation in another clinical trial.
12. Female patients of childbearing potential with a positive pregnancy test, breast feeding, or female patients of childbearing potential without adequate contraception.
13. History and/or presence of drug or alcohol abuse.
14. Patients with psychiatric illness.
15. Irritable bowel syndrome.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-06-18 (Actual); Primary Completion 2013-05-03 (Actual); Study Completion 2013-05-03 (Actual)

PRIMARY OUTCOMES:
AUC of Patients' assessment of gastrointestinal symptoms evaluated by a daily measured VAS scale. | Up to 28 days
  Area under the curve (AUC) of patients' assessment of gastrointestinal symptoms evaluated by daily visual analogue scale (VAS)

SECONDARY OUTCOMES:
Global Subject Outcome Assessment at visit 5 | At day 28 (visit 5)
  Assessed by Global Improvement Scale (substantially worsened/moderately worsened/ marginally worsened/not changed/ marginally improved/ moderately improved/ substantially improved).
Change of the Gastrointestinal Symptoms Profile (GIS) from baseline (visit 3) at the end of study (day 28) | At baseline and day 28
  The GIS is a symptom related score, validated in German language, which allows the investigator to assess the dyspeptic symptoms by asking the patient for the following 10 items (GIS): epigastric pain / upper abdominal pain, abdominal cramps, fullness, early satiety, loss of appetite, sickness, nausea, vomiting, retrosternal discomfort and acid eructation/heartburn. The total GIS score is 40 points and an increasing summary score therefore represents a higher intensity of dyspeptic symptoms.
AUC of reflux symptoms assessment measured by daily VAS scale | Up to 28 days
  Area under the curve (AUC) of assessment of reflux symptoms evaluated by daily visual analogue scale (VAS). VAS is an s an unmarked scale on a line 100 mm in length, indicating from 0 mm (no symptoms) to 100 mm (severe symptoms)
Quality of Life evaluation as assessed by Functional Dyspepsia Quality of Life (FDDQL) | At baseline and day 28
  The FDDQL provided a profile with eight subscores (daily activities, anxiety, diet, sleep, discomfort, health perceptions, coping with disease and impact of stress) as well as a global score. Sub-scale scores and the global score were transformed to a range from "0 = Poor QoL" to "100= Good QoL".
Relative time with an esophageal pH < 4 during 24 hours of measurement by Bravo™ pH system | At day -7/ -5 (screening phase) and day 29/30 if applicable
  The Bravo™ pH system is a new, single use, disposable class I catheter free pH monitoring system, which involves the attachment of a miniaturised radiotelemetry pH capsule to the mucosal wall of the esophagus. It simultaneously measures the pH and transmits data to a pager-sized receiver clipped into the subject's belt
Relative time with an esophageal pH < 4 during 24 hours of measurement using intraluminal impedance | At day -1 (screening phase) and day 29/30 if applicable
  pH measured by pH-metry
Calculation of the DeMeester Score measured based on Bravo™ pH system | At day -7/ -5 (screening phase) and day 29/30 if applicable
  The score is calculated from the following parameters: percentual part of measurement with pH<4, number of reflux periods with a duration of more than 5 minutes, duration of the longest reflux period and total number of reflux periods
System index measurement in parallel to the pH measurement by Bravo™ pH system | At day -7/ -5 (screening phase) and day 29/30 if applicable
  The study patients will be instructed to enter concomitant symptoms (heartburn and upper abdominal pain) which might occur during the measurement by pushing pre-programmed buttons on the data logger A positive symptom index is defined with >50% (more than a half of the concomitant symptoms occur within 5 minutes after bolus exposition)
Calculation of the DeMeester Score based on intraluminal impedance | At day -1 (screening phase) and day 29/30 if applicable
  The score is calculated from the following parameters: percentual part of measurement with pH<4, number of reflux periods with a duration of more than 5 minutes, duration of the longest reflux period and total number of reflux periods)
Bolus exposition time in minutes and as percentual part of measurement time for acid reflux, non-acid reflux and total (acid and non-acid) reflux using intraluminal impedance | At day -1 (screening phase) and day 29/30 if applicable
  Impedance is a measure of the total resistance to current flow between adjacent electrodes. As reflux contents are characterized by different conductivity, which is the inverse of impedance, a pH-independent accurate and practical qualitative analysis of refluxate is possible
Symptom index measurement in parallel to the pH measurement by intraluminal impedance | At day -1 (screening phase) and day 29/30 if applicable
  The study patients will be instructed to enter concomitant symptoms (heartburn, retrosternal discomfort, upper abdominal pain) which might occur during the measurement by pushing pre-programmed buttons on the data logger. A positive symptom index is defined with >50% (more than a half of the concomitant symptoms occur within 5 minutes after bolus exposition).
Global assessment of efficacy judged by patient using a five point Likert scale | At day 28
  1 = very good, 2 = good, 3 = moderate, 4 = poor, 5 = very poor
Global assessment of efficacy judged by physician using a five point Likert scale | At day 28
  1 = very good, 2 = good, 3 = moderate, 4 = poor, 5 = very poor
Change of Individual symptom score from baseline at the end of study (day 28) | At baseline and day 28
  The GIS sub-scores for epigastric pain (item 1) and reflux symptoms (item 10). The sub-scores were assessed and analysed using the following scores: 0 = No problem, 1 = Mild problem, 2 = Moderate problem, 3 = Severe problem, 4 = Very severe

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/